CLINICAL TRIAL: NCT01881997
Title: Randomized Controlled Trial of the Use of Intramuscular Fentanyl for the Incision and Drainage of Abscess in the Emergency Department
Brief Title: Pain Management in ED for Incision and Drainage of Abscess
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB modifications made study impractical.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Larry J. Baraff, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-001068
Record Dates: First submitted 2011-04-01; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Abscess
Keywords: Procedure; Abscess; Emergency Department; Opioid; Fentanyl
MeSH Terms: conditions — Abscess; Emergencies | interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): IM normal saline
  Interventions: Drug: Normal Saline
- Fentanyl (Experimental): IM Fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl Intramuscular (IM), 1ugm/kg, x1
  Arms: Fentanyl
Drug: Normal Saline — IM normal saline
  Arms: Normal Saline

SUMMARY:
Patients presenting with painful procedures in the Emergency Department (ED) have been shown to frequently have inadequate pain management. The incision and drainage (I&D) of an abscess is a common procedure that is viewed by many emergency physicians as only requiring a localized anesthetic for pain management. However, it has been documented in previous research that there can be disconnect between what emergency medicine physicians interpret as painful and what patients experience as pain. A trial will be conducted to focus on use of intramuscular (IM) Fentanyl as an intervention to help alleviate pain associated with the incision and drainage of an abscess. This is a procedure that rarely receives systemic opioids.

This double blinded protocol will randomize a total of 50 patients patients with abscesses to receive either a combination of Fentanyl IM followed by subcutaneous (SC) local bupivicaine analgesia or Normal Saline IM followed by SC local bupivicaine analgesia. Only opiate naive patients will be enrolled. The primary outcomes studied are patients overall satisfaction with procedure, and patients level of pain associated with the procedure.

DETAILED DESCRIPTION:
Patients presenting with painful procedures in the Emergency Department (ED) have been shown to frequently have inadequate pain management. The incision and drainage of an abscess is a common procedure that is usually treated by emergency physicians with only localized anesthetic for pain management. For those abscesses that require incision and drainage, a physician will usually inject a local anesthetic to help decrease sensation to the affected area prior to incision and drainage. Occasionally, physicians will administer a systemic pain medication, in addition to the localized anesthetic, as a method to better help alleviate pain associated with more complex procedures.

Wilson and Pendleton (1989) wrote a landmark study that highlighted the problem of physicians undertreating patients pain in the ED, a problem known as oligoanalgesia. They found that only 50% of patients with moderate to severe pain were receiving narcotics. Since then the literature has highlighted a number of additional deficits in the use of pain medication in the ED to include the amount of time it takes patients to receive medication, the lack of education medical personnel receive in pain management, the bias that physicians have toward using pain medication, and the lack of pain medication given for painful procedures. Five areas of inadequate management of painful conditions in the ED include 1) failure to acknowledge pain, 2) failure to assess initial pain, 3) failure to have pain management guidelines, 4) failure to document pain and assess treatment adequacy, and 5) failure to meet patients expectations. The use of adequate pain medication for painful procedures covers has been a recent attempt to fill in the gap of one area contributing to oligoanalgesia.

Incision and drainage procedures are a common condition that emergency physicians manage yet there is no evidence to suggest whether they are appropriately managing the pain associated with their treatment. We propose a trial to determine whether intramuscular (IM) Fentanyl, given prior to the incision and drainage of the abscess, decreases the level of pain during/after the procedure and increases the patients overall satisfaction with the procedure.

This double blind protocol will randomize 50 patients with abscesses to receive either a combination of an intramuscular injection of Fentanyl followed by subcutaneous (SC) local bupivacaine analgesia (Fentanyl Group), or a combination of an intramuscular injection of normal saline (Control Group) IM followed by SC local bupivacaine analgesia. Patients will receive a questioner administered by a research assistant after the procedure to assess outcomes of study.

Neither treating physicians, nurses nor patients and research assistants will be aware to which group the patient has been randomized. Fentanyl was chosen due to the rapidity of onset (7-8 minutes) and clearance (1-2 hours). The choice of abscess was made given the ease at which to make a diagnosis, standard treatment with incision and drainage and known association with pain during and after the procedure.

After appropriate identification, screening, and consenting, the patient will then be randomized to receive intramuscular Fentanyl (1 ug/kg) OR Normal Saline (1.5 ml) 7-8 minutes before the procedure is began. Patients in either group will still receive usual care with local subcutaneous bupivacaine anesthetics. Patients are at liberty to request more local subcutaneous bupivacaine and or more pain systemic pain medication and the treating provider may deliver more at their discretion. Contamination may occur if patients receiving IM Normal Saline request systemic narcotics for pain levels not controlled with local bupivacaine alone. These patients may receive systemic narcotics again at the discretion of treating providers. However all patients will remain in the initial group to which they were assigned and data will be evaluated on an intention to treat analysis basis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and < 65 years
* Presenting with a simple abscesses requiring incision and drainage
* Treating physician has to state that the patient's usual treatment would not include systemic opioids before incision and drainage.

Exclusion Criteria:

* Patients are unable to consent to procedure the procedure
* Patients are less than age 18 or older than age 65
* Patients are unable to avoid driving for 2 hours after administration of the intramuscular medication (Fentanyl or placebo)
* Patients have hypersensitivity or allergy to Fentanyl
* Patients are pregnant
* Patients have taken a narcotic pain medication in the last 14 days
* Patients have a history of drug or alcohol addiction
* Patients have taken an monoamine oxidase (MAO) inhibitor in the last 14 days (such as furazolidone (Furoxone), isocarboxazid (Marplan), phenelzine (Nardil), rasagiline (Azilect), selegiline (Eldepryl, Emsam, Zelapar), or tranylcypromine (Parnate)
* Patients have a breathing disorder such as chronic obstructive pulmonary disease
* Patients have a history of head injury or brain tumor
* Patients have a heart rhythm disorder
* Patients have seizures or epilepsy
* Patients have mental illness such as depression, hallucinations
* Patients have low blood pressure
* Patients have liver or kidney disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Highest level of pain during the incision and drainage of the abscess | Participants will be followed for the duration of hospital stay
  After the procedure the following question will be asked via a survey:
  On a scale of 1-10 with 10 being the worst possible pain, what was your highest level of pain during the incision and drainage of the abscess? The answer will be collected via a visual analog scale.
Safety of Intramuscular Injection of Fentanyl | Participants will be followed for the duration of hospital stay
  All patients will be monitored to see if any of the following occur after administration of Fentanyl:
  Adverse effects
  * decreased oxygen saturation <95%
  * respiratory depression
  * bradycardia
  * hypotension
  * anaphylaxis or laryngospasm or bronchoconstriction
  * muscle rigidity
  * other:
  Side effects
  * nausea
  * itching
  * drowsiness
  Treatment needed
  * O2
  * IV Fluids
  * Medications: Specify name and dose
  * Other, specify:

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Baraff, MD, Principal Investigator — University of California, Los Angeles; Joshua W Elder, B.S., Study Director — University of California, Los Angeles; Adaira Landry, B.A., Study Director — University of California, Los Angeles

REFERENCES:
- [Result] Wilson JE, Pendleton JM. Oligoanalgesia in the emergency department. Am J Emerg Med. 1989 Nov;7(6):620-3. doi: 10.1016/0735-6757(89)90286-6. PMID 2803357
- [Result] Fosnocht DE, Swanson ER, Bossart P. Patient expectations for pain medication delivery. Am J Emerg Med. 2001 Sep;19(5):399-402. doi: 10.1053/ajem.2001.24462. PMID 11555797
- [Result] Motov SM, Khan AN. Problems and barriers of pain management in the emergency department: Are we ever going to get better? J Pain Res. 2008 Dec 9;2:5-11. PMID 21197290
- [Result] Downey LV, Zun LS. Pain management in the emergency department and its relationship to patient satisfaction. J Emerg Trauma Shock. 2010 Oct;3(4):326-30. doi: 10.4103/0974-2700.70749. PMID 21063553
- [Result] Yanuka M, Soffer D, Halpern P. An interventional study to improve the quality of analgesia in the emergency department. CJEM. 2008 Sep;10(5):435-9. doi: 10.1017/s1481803500010526. PMID 18826731
- [Result] Fry M, Holdgate A. Nurse-initiated intravenous morphine in the emergency department: efficacy, rate of adverse events and impact on time to analgesia. Emerg Med (Fremantle). 2002 Sep;14(3):249-54. doi: 10.1046/j.1442-2026.2002.00339.x. PMID 12487041
- [Result] Schechter NL, Weisman SJ, Rosenblum M, Bernstein B, Conard PL. The use of oral transmucosal fentanyl citrate for painful procedures in children. Pediatrics. 1995 Mar;95(3):335-9. PMID 7862469
- [Result] Weisman SJ, Bernstein B, Schechter NL. Consequences of inadequate analgesia during painful procedures in children. Arch Pediatr Adolesc Med. 1998 Feb;152(2):147-9. doi: 10.1001/archpedi.152.2.147. PMID 9491040
- [Result] O'Malley GF, Dominici P, Giraldo P, Aguilera E, Verma M, Lares C, Burger P, Williams E. Routine packing of simple cutaneous abscesses is painful and probably unnecessary. Acad Emerg Med. 2009 May;16(5):470-3. doi: 10.1111/j.1553-2712.2009.00409.x. Epub 2009 Apr 10. PMID 19388915
- [Result] Curtis KM, Henriques HF, Fanciullo G, Reynolds CM, Suber F. A fentanyl-based pain management protocol provides early analgesia for adult trauma patients. J Trauma. 2007 Oct;63(4):819-26. doi: 10.1097/01.ta.0000240979.31046.98. PMID 18090011